CLINICAL TRIAL: NCT05066594
Title: Observational Registry of Transoral Incisionless Fundoplication (Creation of a New Gastroesophageal Valve) in Patients With Gastroesophageal Reflux Disease
Brief Title: Observational Registry of Transoral Incisionless Fundoplication (TIF) for Gastroesophageal Reflux Disease (GERD)
Acronym: TIF/2021
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Pier Alberto Testoni, Head of Gastroenterology and Digestive Endoscopy, IRCCS San Raffaele
Other Study IDs: TIF REGISTRY 2021
Record Dates: First submitted 2021-04-29; First posted 2021-10-04 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-09

CONDITIONS: Gastro Esophageal Reflux
Keywords: Fundoplication; Endoscopy, Digestive System; Gastro Esophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Transoral incisionless fundoplication with EsophyX device (EndoGastric Solutions): Patients treated by transoral incisionless fundoplication (TIF) using the EsophyX device (EndoGastric Solutions) for gastro-esophageal reflux disease will be enrolled in the registry and clinically followed-up for 5 years from the date of TIF procedure.
  Interventions: Device: Transoral incisionless fundoplication

INTERVENTIONS:
Device: Transoral incisionless fundoplication — The intervention of transoral incisionless fundoplication using the EsophyX (EndoGastric Solutions) system allows, through the endoscopic route, the creation of a cardial neovalve of approximately 270 ° by placing 20-28 polyethylene sutures on the cardial circumference, resulting in an anti-reflux plastic functionally similar to that obtained with the surgical fundoplication.

SUMMARY:
This observational registry aims to: 1) record the TIF interventions in patients with esophageal or extra-esophageal symptoms; 2) to monitor the therapy response through the clinical experience in terms of effect on the use and dosage of proton pump inhibitors (PPIs) and on the GERD-Health Related Quality of Life (HRQL) and Reflux Symptom Index (RSI) questionnaires scores; 3) to characterize the treated patients population and the predictive factors of TIF success, identifying the subpopulation who may effectively benefit from TIF.

DETAILED DESCRIPTION:
After being evaluated according to the clinical indication for the treatment of symptomatic gastro-esophageal reflux disease (GERD with esophageal or extraesophageal symptoms) by transoral incisionless fundoplication (TIF) and, thus, being treated by TIF using the EsophyX device, all patients giving specific informed consent will enter a 3-year enrollment registry with a 5-year follow-up for each patient through post-TIF routine practice visits and examinations.

ELIGIBILITY:
Inclusion Criteria for enrollment:

* Clinical indication to undergo transoral incisionless fundoplication (TIF) with the EsophyX device for treatment of chronic gastro-esophageal reflux disease;
* Availability for prolonged follow-up (5 years) after TIF at San Raffaele Hospital;
* Signed informed consent for participation in the observational registry.

Exclusion Criteria for enrollment:

* Absence of clinical indication to undergo transoral incisionless fundoplication (TIF) with the EsophyX device for treatment of chronic gastro-esophageal reflux disease;
* Unavailability for prolonged follow-up (5 years) after TIF at San Raffaele Hospital;
* No signed informed consent for participation in the observational registry.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion criteria for TIF: >12 months esophageal or extraesophageal symptoms from gastroesophageal reflux, despite >6 months therapy with PPI; cardial valve Hill's degree >III; pathological gastroesophageal reflux; hiatal hernia ≤2 cm.
  Exclusion criteria for TIF: hiatal hernia >2 cm; paraesophageal hernia; severe esophageal motility disorder or Los Angeles grade C and D esophagitis; esophageal stenosis, diverticula, infections; pregnancy, breastfeeding; bleeding disorders; malignant neoplasm; immunosuppressant therapy; portal hypertension; esophageal varices; eosinophilic esophagitis; autoimmune esophagitis; BMI ≥35; limited mobility of the neck; patients for whom the use of the EsophyX device is contraindicated.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Medical use and dosage | Yearly, up to 5 years from the date of the intervention
  Need to use proton pump inhibitors (PPI), and at what dosage, to control the gastro-esophageal reflux symptoms after intervention

SECONDARY OUTCOMES:
Health Related Quality of Life questionnaire score | Yearly, up to 5 years from the date of the intervention
  Modification of the scores from the gastro-esophageal reflux disease-health related quality of life (GERD-HRQL) questionnaire (off proton pump inhibitors), according to a Likert scale from 0 (absence of symptoms) to 5 (symptoms do not allow for normal daily activity), after intervention compared with baseline
Reflux Symptom Index questionnaire score | Yearly, up to 5 years from the date of the intervention
  Modification of the scores from the reflux symptom index (GERD-RSI) questionnaire (off proton pump inhibitors), according to a Likert scale from 0 (no problem) to 5 (severe problem) after the intervention compared with baseline
Esophagitis | 6 months and 12 months after the date of the intervention
  Presence and degree of esophagitis according to the Los Angeles classification (grade A, grade B, grade C, grade D) after the intervention
Hill's grade of the gastro-esophageal flap valve | 6 months and 12 months after the date of the intervention
  Degree of continence of the neo gastro-esophageal flap valve according to the Hill classification (grade I, grade II, grade III, grade IV) after the intervention
Jobe's length of the gastro-esophageal valve | 6 months and 12 months after the date of the intervention
  Length of the fold of the neo gastro-esophageal valve according to the criteria of Jobe et al. after the intervention
Barrett's esophagus | 6 months and 12 months after the date of the intervention
  Presence and degree of Barrett's esophagus according to the Prague classification (C, M) after the intervention
High-resolution esophageal manometry findings | 12 months after the date of the intervention
  Esophageal manometry measurements after the intervention
24-hour esophageal pH-metry findings | 12 months and 24 months after the date of the intervention
  24-hour esophageal pH-metry measurements off proton pump inhibitors after the intervention
24-hour esophageal impedancemetry findings | 12 months and 24 months after the date of the intervention
  24-hour esophageal pH-impedance measurements off proton pump inhibitors after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Pier Alberto Testoni, Prof., Principal Investigator — IRCCS San Raffaele
Locations (1):
- IRCCS San Raffaele, Milan, Italy